CLINICAL TRIAL: NCT07333898
Title: Digital Measurements of Motor and Voice Functions in FTD
Status: Not yet recruiting | Type: Observational
Sponsor: BioSensics (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: BioDigit FTLD-03; Digital Assessment Tools Award (Other Grant/Funding Number: AFTD)
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Frontotemporal Lobar Degeneration (FTLD); Frontotemporal Dementia (FTD); Corticobasal Syndrome; Corticobasal Syndrome(CBS); Corticobasal Degeneration
Keywords: digital health; wearable sensors; frontotemporal lobar degeneration
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Frontotemporal Dementia; Corticobasal Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frontotemporal Lobar Degeneration (FTLD): 20 patients who have a clinical diagnosis of possible or probable FTLD syndrome phenotype.

SUMMARY:
The primary objective of this clinical study is to provide the initial validation for monitoring biomarkers of symptoms and functioning for individuals with FTLD syndromes.

Researchers at BioSensics and Johns Hopkins School of Medicine will use wearable sensors, computerized speech, psychomotor, and cognitive assessments to create outcome measures and digital biomarkers for FTLD syndromes. Researchers will deploy this digital health solution to monitor 20 patients with FTLD syndromes for 12 months with study visits every 3 months.

DETAILED DESCRIPTION:
Frontotemporal degeneration (FTD) spans the spectrum of rare neurodegenerative disorders affecting movement, behavior, and cognitive function. FTD represents a group of disorders including progressive supranuclear palsy (PSP - a severe and rapidly progressive FTD disorder estimated to affect at least 20,000 Americans), frontotemporal dementia (FTD, the second most common cause of early-onset (<65) dementia), primary progressive aphasia, semantic dementia, and corticobasal syndrome.

The primary objective of this clinical study is to provide the initial validation for monitoring biomarkers of symptoms and functioning for individuals with FTLD syndromes.

Twenty patients with FTLD syndromes will be recruited from Johns Hopkins University School of medicine to participate in this 12-month study with visits every 3 months. The investigators aim to assess the correlation between outcomes as measured by the PAMSys pendant and PAMSys ULM wrist monitoring sensors, and clinical/functional assessments used for FTLD syndromes (bvFTD, nfPPA, SD, and CBS), including the FTD Rating Scale (FTDRS), Cortical Basal ganglia Functional Scale (CBFS), PSP Rating Scale (PSPRS), Frontal Assessment Battery (FAB) (lexical fluency and Go-No-Go tasks), FTLD-CDR, modified Interpersonal Reactivity Index (mIRI Perspective Taking and Empathic Concern subscales summed to obtain a total Empathy score), the Pyramids and Palm Trees test (PPT), the Bedside Western Aphasia Battery-Revised (BWAB-R), digit span, phonemic fluency, category fluency, color trails, and trails A and B in individuals with different stages of FTLD disease severity. The results will be used to develop and validate monitoring symptoms and function in FTLD syndromes. In an exploratory aim, the caregiver burden (Zarit Burden Inventory) and its relationship to patients' empathy levels (mIRI) will be assessed.

The secondary objective of this study is to conduct free-flowing interviews with participants and clinical experts using the Technology Acceptance Model (TAM). This approach will help us examine perceptions of benefit, technology acceptance, technological anxiety, trust, facilitating conditions, perceived risk, and attitudes towards use from the perspectives of both patients and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 40 years or older with a clinical diagnosis of possible or probable FTLD syndrome phenotype.
* Participants must be fluent in reading and speaking English and must be capable of providing informed consent based on the principal investigator's judgment.
* Individuals eligible for inclusion must be able to comply with the protocol per the investigator's judgment and must have a caregiver or study partner who is willing and able to assist with all study-related procedures.

Exclusion Criteria:

* Any neurological, medical, or psychiatric condition that would preclude or confound participation in study activities based on the investigator's judgment.
* Individuals who have a history of frequent falls defined as more than 5 falls per month.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study intends to enroll a diverse population of individuals representative of the general FTLD syndrome population. There are no restrictions based on race or ethnic origin. This study will enroll both male and female participants aged 40 years or older with a clinical diagnosis of possible or probable FTLD syndrome phenotype.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Monitoring | 12 months
  Following each clinical visit, participants will be asked to wear a PAMSys pendant sensor and two PAMSys ULM wrist sensors for 14 days at home. The average daily number of steps will be measured using the PAMSys pendant.
Hand Function Monitoring | 12 months
  Following each clinical visit, participants will be asked to wear two PAMSys ULM wrist sensors for 14 days at home. Average daily number of hand goal-directed movements will be measured using the PAMSys ULM wrist sensors.

SECONDARY OUTCOMES:
Zarit Burden Interview (ZBI) | 12 months
  The ZBI is completed by a reliable caregiver. The ZBI scores range from 0-88, where 88 represents a worse outcome.
Montreal Cognitive Assessment (MoCA) | 12 months
  This is a brief global cognitive screening assessment. Scores range from 0 to 30 where 0 represents a worse outcome.
Frontal Assessment Battery (FAB) | 12 months
  This is a short screening tool that measures executive functions to help differentiate between types of dementia or assess frontal lobe dysfunction. It consists of six subtests that evaluate a person's conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy, with a maximum score of 18. The FAB is a quick and simple test, with each subtest scored from 0 to 3.
Cortical Basal Ganglia Functional Scale (CBFS) | 12 months
  The CBFS is a rating scale that evaluates experiences in daily living (EDL's) and consists of 14 questions on Motor EDL's and 17 questions on Non-Motor EDL's, each of which are rated on a Likert 5 point scale rating function from 0 to 4, where 0 = Normal or No problems and 4 = Severe problems. The questions are for the patient, but should be answered by both the patient and their caregiver together.
Progressive Supranuclear Palsy Rating Scale (PSPRS) | 12 months
  The PSP Rating Scale (PSPRS) is a 28-item clinical assessment used to measure the severity and progression of Progressive Supranuclear Palsy (PSP). Out of the 28-items, 6 are scored on a 3 point scale (0-3) and 22 are scored on a 4 point scale (0-4). The PSPRS ranges from a score of 0-100 with a higher number representing a greater impairment from the disease.

OTHER OUTCOMES:
Digital Speech Assessment | 12 months
  Using a study tablet, participants will perform a series of digital speech assessments. The collected speech data will be analyzed using BioDigit Speech, an automatic speech analysis software developed by BioSensics.
Digital Cognitive Assessment | 12 months
  Using a study tablet, participants will perform a series of digital cognitive assessments.
Digital Fine Motor Control Assessment | 12 months
  Using a study tablet, participants will perform a series of tapping tests.